CLINICAL TRIAL: NCT03264040
Title: Biomarker for Mannosidosis Disease - An International, Multicenter, Epidemiological Protocol
Brief Title: Biomarker for Mannosidosis Disease (BioMannosidosis)
Acronym: BioMannosido
Status: Withdrawn | Type: Observational
Why Stopped: Transition to BioMetabol
Sponsor: CENTOGENE GmbH Rostock (Industry)
Responsible Party: Sponsor
Other Study IDs: BMA 06-2018
Record Dates: First submitted 2017-08-24; First posted 2017-08-28 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Alpha-Mannosidase B Deficiency; Lysosomal Alpha B Mannosidosis; Alpha-Mannosidase Deficiency
Keywords: Mannosidosis; Biomarker
MeSH Terms: conditions — alpha-Mannosidosis; Mannosidase Deficiency Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — For the development of the new biomarkers using the technique of Mass-spectrometry 2,7 ml EDTA blood or a dry blood spot filter card are taken. To proof the correct Mannosidosis diagnosis in those patients where up to the en-rollment in the study no genetic testing has been done, sequencing of Manno-sidosis disease will be done.
  The analyses will be done at the Centogene AG Am Strande 7 18055 Rostock Germany
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observation: Patients with Mannosidosis disease or high-grade suspicion for Mannosidosis disease

SUMMARY:
Development of a new MS-based biomarker for the early and sensitive diagnosis of Mannosidosis disease from blood (plasma)

DETAILED DESCRIPTION:
Alpha-Mannosidosis is a rare lysosomal storage disorder of the Glycoprotein family of diseases and is closely related to Mucopolysaccharidoses.

Alpha-Mannosidosis was first described by Dr Oekerman, from Lund in Sweden in 1967. There is another variant known as Beta-Mannosidosis, which is extremely rare and has produced a wide range of clinical abnormalities in the few patients described with this disorder.

A Alpha-Mannosidosis is a rare inherited disorder that causes problems in many organs and tissues of the body. Affected individuals may have intellectual disability, distinctive facial features, and skeletal abnormalities. Characteristic facial features can include a large head, prominent forehead, low hairline, rounded eyebrows, large ears, flattened bridge of the nose, protruding jaw, widely spaced teeth, overgrown gums, and large tongue. The skeletal abnormalities that can occur in this disorder include reduced bone density (osteopenia), thickening of the bones at the top of the skull (calvaria), deformations of the bones in the spine (vertebrae), bowed legs or knock knees, and deterioration of the bones and joints.

Affected individuals may also experience difficulty in coordinating movements (ataxia); muscle weakness (myopathy); delay in developing motor skills such as sitting and walking; speech impairments; increased risk of infections; enlargement of the liver and spleen (hepatosplenomegaly); a buildup of fluid in the brain (hydrocepha-lus); hearing loss; and a clouding of the lens of the eye (cataract). Some people with Alpha-Mannosidosis experience psychiatric symptoms such as depression, anxiety, or hallucinations; episodes of psychiatric disturbance may be triggered by stressors such as having undergone surgery, emotional upset, or changes in routine.

The signs and symptoms of Alpha-Mannosidosis can range from mild to severe. The disorder may appear in infancy with rapid progression and severe neurological deterioration. Individuals with this early-onset form of Alpha-Mannosidosis often do not survive past childhood. In the most severe cases, an affected fetus may die before birth. Other individuals with Alpha-Mannosidosis experience milder signs and symptoms that appear later and progress more slowly. People with later-onset alpha-mannosidosis may survive into their fifties. The mildest cases may be detected only through laboratory testing and result in few if any symptoms.

Alpha-mannosidosis is estimated to occur in approximately 1 in 500,000 people worldwide.

Mutations in the MAN2B1 gene cause Alpha-Mannosidosis. This gene provides instructions for making the enzyme alpha-mannosidase. This enzyme works in the lysosomes, which are compartments that digest and recycle materials in the cell. With-in lysosomes, the enzyme helps break down complexes of sugar molecules (oligo-saccharides) attached to certain proteins (glycoproteins). In particular, alpha-mannosidase helps break down oligosaccharides containing a sugar molecule called mannose.

Mutations in the MAN2B1 gene interfere with the ability of the alpha-mannosidase enzyme to perform its role in breaking down mannose-containing oligosaccharides. These oligosaccharides accumulate in the lysosomes and cause cells to malfunction and eventually die. Tissues and organs are damaged by the abnormal accumulation of oligosaccharides and the resulting cell death, leading to the characteristic features of Alpha-Mannosidosis.

New methods, like mass-spectrometry give a good chance to characterize specific metabolic alterations in the blood (plasma) of affected patients that allow diagnosing in the future the disease earlier, with a higher sensitivity and specificity.

Therefore it is the goal of the study to identify and validate a new biochemical marker from the plasma of the affected patients helping to benefit other patients by an early diagnose and thereby with an earlier treatment.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent will be obtained from the patient or the parents before any study related procedures.
* Patients of both genders older than 2 months
* The patient has a diagnosis of Alpha-Mannosidosis disease or a high grade suspicion for Alpha-Mannosidosis disease
* High grade suspicion present, if one or more inclusion criteria are valid:

  * Positive family anamnesis for Alpha-Mannosidosis disease
  * rounded eyebrows
  * large head
  * large ears
  * flattened bridge of the nose
  * deformations of the bones in the spine (vertebrae)

Exclusion Criteria:

* No Informed consent from the patient or the parents before any study related procedures.
* Patients of both gender younger than 2 months
* No diagnosis of Alpha-Mannosidosis disease or no valid criteria for profound suspicion of Alpha-Mannosidosis disease

Min Age: 2 Months | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Mannosidosis disease or high-grade suspicion for Mannosidosis disease
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Development of a new MS-based biomarker for the early and sensitive diagno-sis of Mannosidosis disease from blood (plasma) | 24 months
  New methods, like mass-spectrometry give a good chance to characterize specific metabolic alterations in the blood of affected patients that allow diagnosing in the future the disease earlier, with a higher sensitivity and specificity.

SECONDARY OUTCOMES:
Testing for clinical robustness, specificity and long-term stability of the bi-omarker | 36 months
  the goal of the study to identify and validate a new biochemical marker from the blood of the affected patients helping to benefit other patients by an early diagnose and thereby with an earlier treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Bauer, Prof., Study Chair — Centogene GmbH
Locations (3):
- Centogene GmbH, Rostock, Germany
- Navi Mumbai Institute of Research In Mental And Neurological Handicap (NIRMAN), Mumbai, India
- Lady Ridgeway Hospital for Children, Colombo, Sri Lanka